CLINICAL TRIAL: NCT02742285
Title: Comparison of Lumefantrine Concentrations Measured in Venous Plasma Versus in Dried Capillary Blood Spot Samples in Healthy Volunteers.
Brief Title: Lumefantrine in Venous Plasma Versus Dried Capillary Blood Spot
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Thierry Buclin (Other)
Responsible Party: Sponsor-Investigator, Thierry Buclin, Professor, Centre Hospitalier Universitaire Vaudois
Organization: Centre Hospitalier Universitaire Vaudois (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DBS-ALU
Record Dates: First submitted 2016-04-01; First posted 2016-04-19 (Estimated); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: Malaria
Keywords: antimalarials; blood samples; drug concentrations; pharmacokinetics; lumefantrine; healthy volunteers
MeSH Terms: conditions — Malaria | interventions — Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Artemether + lumefantrine (Other): One single adult dose of artemether + lumefantrine 80 + 480 mg
  Interventions: Drug: Artemether + lumefantrine

INTERVENTIONS:
Drug: Artemether + lumefantrine — A single adult dose of artemether-lumefantrine will be administered on a unique occasion together with food. Venous and capillary blood samples will be collected at 6 to 10 time points, as defined before drug administration with each volunteer.
  Other Names: (Riamet)

SUMMARY:
Measurement of the concentration of antimalarials in the blood of the general population helps estimating the overall drug pressure and is used in efficacy studies. The current sampling standard for drug measurement is plasma obtained by venous puncture. The use of a Dried Blood Spots (DBS) sampling strategy can make some aspects of field trials conditions easier, but concordance with usual venous sampling is not yet established.

The current work will allow validating the concentrations of lumefantrine measured in the DBS samples collected during the field trials and validate the use of DBS for future studies. In addition, bearing in mind the substantial deployment of artemether-lumefantrine combinations supplies throughout most malaria endemic countries, this study may improve our understanding of lumefantrine and artemether distribution in the blood compartments and generate knowledge for further developing analytical methods for drug measurement.

The overall purpose of this study is to validate the dried blood spots as a sampling method for the analysis of lumefantrine.

The primary objective is to assess the concordance between lumefantrine plasma and dried blood spots (DBS) concentrations.

The investigators also aim at describing lumefantrine's distribution in the different blood compartments: binding to plasma proteins, total in plasma, inside the red blood cells, total in whole blood.

DETAILED DESCRIPTION:
(Details available on request)

ELIGIBILITY:
Inclusion Criteria:

* Absence of current drug treatment (except hormonal contraception, an additional barrier method is strongly advised)
* 12-lead ECG without significant abnormalities
* The subject understands the procedures, agrees to participate and is willing to give written informed consent
* The subject agrees to be available for at least 5 blood sampling after drug administration, at scheduled time points.

Exclusion Criteria:

* History of any major medical disorder
* Any recent acute illness which could expose the subject to a higher risk or might confound the results of the study
* Current pregnancy or breast-feeding
* Congenital prolongation of the QT interval (e.g., long QT syndrome) or any other clinical condition known to prolong the corrected QT interval
* Family history of congenital prolongation of the QT interval or sudden death
* Known disturbances of electrolyte balance
* Known liver disorder of any type, even if no medical treatment is needed. Gilbert syndrome will be tolerated, if mild
* Treatment in the previous three months with any drug known to have well-defined potential for toxicity to a major organ
* History of hypersensitivity to any component of the drug
* History of hypersensitivity to any drug if considered as serious
* History of alcohol or drug abuse
* Present consumption of a large quantity of alcohol or wine (>0.5 L wine/day) or equivalent. Consumption of reasonable amount of wine (0.3 L) or of beer is acceptable, except between Day -1 to Day 3 of drug administration
* Use of any medication the week prior to study or as based on 5 plasma half-life rule and up to 48 hours post drug administration
* Participation in a clinical trial in the previous 3 months unless no treatment provided and low amount of blood collected
* Occupation which might interfere with visits and blood sampling during the study
* Psychological status which could have an impact on subject's ability to give informed consent
* Any feature of subject's medical history or present condition which, in the investigator's opinion, could confound the results of the study, complicate their interpretation or represent a potential risk for the subject

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2016-05; Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Concordance of concentrations of lumefantrine measured in dried capillary blood spot samples (DBS) and in plasma, at different time-points after the administration of a single oral adult dose of artemether-lumefantrine. | Within the first two weeks after drug intake

SECONDARY OUTCOMES:
Concordance of concentrations of desbutyl-lumefantrine measured in DBS and in plasma | Within the first two weeks after drug intake
Concordance of lumefantrine and desbutyl-lumefantrine concentrations measured in dried venous blood spot samples and in plasma | Within the first two weeks after drug intake
Concordance of concentration of lumefantrine and desbutyl-lumefantrine measured in whole venous blood and in plasma | Within the first two weeks after drug intake
Determination of a ratio of intra-erythrocyte and plasma concentrations of lumefantrine and desbutyl-lumefantrine over time (corrected for hematocrit) | Within the first two weeks after drug intake
Determination of a ratio of unbound plasma concentration and total plasma concentration of lumefantrine and desbutyl-lumefantrine over time | Within the first two weeks after drug intake
Determination of the limit of quantification of artemether and dihydroartemisinin in dried blood spots samples, using the standard method of a calibration curve | Within the first 24 hours after drug intake
Determination the relative precision of lumefantrine and desbutyl-lumefantrine concentrations in dried blood spots versus in plasma, using triplicate measurements and a hierarchical non-linear regression model | Within the first two weeks after drug intake

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Buclin, Professor, Principal Investigator — Division of Clinical Pharmacology, University Hospital, Lausanne, Switzerland
Locations (1):
- Division of Clinical Pharmacology, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Yes